CLINICAL TRIAL: NCT05810311
Title: The Effect of Roxadustat on the Levels of Renal Oxygenation in Patients With Diabetes Nephropathy (FOXTROT)
Brief Title: The Effect of Roxadustat on Renal Oxygenation in Diabetes Nephropathy
Acronym: FOXTROT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Region Stockholm (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FOXTROT
Record Dates: First submitted 2023-03-24; First posted 2023-04-12 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Complications; Diabetes; Nephropathy (Manifestation)
Keywords: HIF; Hypoxia; Diabetes mellitus; Nephropathy; BOLD-MRI; Kidney oxygenation
MeSH Terms: conditions — Diabetes Complications; Diabetes Mellitus; Kidney Diseases; Hypoxia | interventions — roxadustat; Darbepoetin alfa

STUDY DESIGN:
Intervention Model Description: The research design is a randomized prospective, open-label study with parallel groups of 15 patients/group with non-dialysis dependent DKD CKD stage 3-4 with Hb <10g/dl.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Roxadustat (Active Comparator): The group will receive Roxadustat (Evrenzo) three times weekly at an initial dose of 70mg (for body weight <100.0 kg) or 100 mg (for body weight weight ≥100.0 kg). The dosage for both arms will be adjusted to keep Hb at the recommended levels between 11-12g/dl.
  Interventions: Drug: Roxadustat
- Darbepoietin alpha (Active Comparator): The control group will receive darbepoietin alpha (Aranesp) s.c. 0.45mg/kg once a week. The dosage for both arms will be adjusted to keep Hb at the recommended levels between 11-12g/dl.
  Interventions: Drug: Darbepoietin Alfa

INTERVENTIONS:
Drug: Roxadustat — The group will receive Roxadustat (Evrenzo) three times weekly at an initial dose of 70mg (for body weight <100.0 kg) or 100 mg (for body weight weight ≥100.0 kg). The dosage for both arms will be adjusted to keep Hb at the recommended levels between 11-12g/dl.
  The aim is to investigate the effects of systemic administration of Evrenzo (Roxadustat [RD]) or Aranesp (darbepoetin alpha [DA]) on the levels of renal oxygenation in patients with diabetic nephropathy and associated anemia.
  Other Names: Evrenzo
  Arms: Roxadustat
Drug: Darbepoietin Alfa — The control group will receive darbepoietin alpha (Aranesp) s.c. 0.45mg/kg once a week. The dosage for both arms will be adjusted to keep Hb at the recommended levels between 11-12g/dl.
  The aim is to investigate the effects of systemic administration of Evrenzo (Roxadustat [RD]) or Aranesp (darbepoetin alpha [DA]) on the levels of renal oxygenation in patients with diabetic nephropathy and associated anemia.
  Other Names: Aranesp
  Arms: Darbepoietin alpha

SUMMARY:
The study will investigate if treatment with Roxadustat improves kidney oxygenation in diabetic patients with nephropathy receiving treatment for renal anemia, compared to patients receiving treatment with darbepoetin alpha.

Participants will be randomized to either treatment, and receive equal care for renal anemia. Kidney oxygenation will be examined before treatment start and after 24 weeks using BOLD-MRI (blood oxygen level-defendant MRI), a non-invasive method available for measurement of tissue oxygenation levels that is comparable with direct invasive measurement of partial oxygen pressure. Blood and urin samples will be collected in connection to these visits. The primary endpoint is the change in medullary and cortical R2* (inversely proportional to the tissue oxygenation content) after 24 weeks. Secondary endpoints will be albuminuria and urinary levels of ROS (evaluated by electron paramagnetic resonance (EPR) spectroscopy with CPH spin probes).

DETAILED DESCRIPTION:
Aims

The general aim of this study is to investigate the effects of systemic administration of Evrenzo (Roxadustat [RD]) or Aranesp (darbepoetin alpha [DA]) on the levels of renal oxygenation in patients with diabetic nephropathy and associated anemia.

The investigation will elucidate if RD, a prolyl-hydroxylase (PHD) inhibitor and subsequent Hypoxia-Inducible Factor 1 (HIF) activator, can reduce renal hypoxia, compared to DA, which lacks effects on HIF.

Background

Diabetes complications represent a huge health problem and concern for modern diabetes therapy, with dramatic consequences for the affected individuals and society.

Diabetic kidney disease (DKD) is the most common cause of end-stage renal disease (ESRD) and accounts for a high morbidity and mortality rate in patients with diabetes. Today, the treatment for DKD focuses on optimizing the patients' metabolic control, blood lipid levels and blood pressure, which unfortunately is optimally achieved in just a restricted portion of patients (1). Thus, there is a great need of identifying novel therapies that could improve or prevent progression DKD.

While hyperglycemia is the major factor contributing to the development of diabetes complications, the role of hypoxia has recently become increasingly evident as another central factor in all diabetes complications (2). Several effects may contribute to the development of hypoxia in diabetes, including deficient blood supply secondary to micro- and macro-vascular disease, poor local oxygen diffusion secondary to local oedema, or as a result of increased oxygen consumption (3, 4, 5, 6).

HIF-1, a heterodimeric transcription factor, is a central regulator of cellular adaptive response to hypoxia (7). HIF consists of two subunits (alpha and beta), both constitutively expressed in mammalian cells. In normoxia, HIF-1alpha is continuously degraded by the ubiquitin-proteasome system because of the oxygen-dependent hydroxylation of two key proline residues catalyzed by a group of enzymes known as prolyl-hydroxylases (PHDs) (7). Upon hypoxia, this degradation pathway is suppressed and HIF-1alpha is stabilized, translocates to the nucleus where it dimerizes with HIF-1beta and induces the expression of more than 800 genes involved in angiogenesis, glycolytic energy metabolism, proliferation and survival that enables the cells to adapt to reduced oxygen availability (8, 9). HIF-1 is central for expression of several angiogenic growth factors (e.g., VEGF, erythropoietin (EPO), stromal cell-derived factor-1alpha) (10).

Lately, accumulating evidence points to a defective cellular response to hypoxia in diabetes. This defective hypoxia response has been shown to be present in all tissues that develop complications in both animal models for diabetes and in patients with diabetes as a consequence of impaired HIF signaling, and there is a direct suppressive effect of hyperglycemia on HIF function (11). Studies in animal models of diabetes have demonstrated that restoring HIF function in hyperglycemia can prevent the development of multiple diabetes complications, including DKD (7).

RD is a PHD inhibitor that stabilizes HIF-1 by preventing PHD dependent degradation of HIF-1alpha, and has recently been approved for treatment of renal anemia. As hypoxia plays a central pathogenic role even in the early stages of DKD (12), and activation of HIF signaling has recently been demonstrated to have protective effects in animal models of DKD (13), it is of great interest to also investigate the potential role of RD as a targeted therapy for DKD in humans.

The presently proposed project aims to investigate the potential of RD to improve renal oxygenation in patients with DKD and anemia, compared to DA which lacks the above-mentioned effects on HIF and is an alternative treatment for the same condition. To examine this the investigators plan to use BOLD-MRI (blood oxygen level-defendant MRI), a non-invasive method available for measurement of tissue oxygenation levels that is comparable with direct invasive measurement of partial oxygen pressure (14).

Research design

The research design is a randomized prospective, open-label study with parallel groups of 15 participants/group with non-dialysis dependent DKD CKD stage 3-4 with Hb <10g/dl (the level of Hb recommended for RD/DA treatment). One group will receive Roxadustat (Evrenzo) three times weekly at an initial dose of 70mg (for body weight <100.0 kg) or 100 mg (for body weight weight ≥100.0 kg). The control group will receive darbepoietin alpha (Aranesp) s.c. 0.45mg/kg once a week. The dosage for both arms will be adjusted to keep Hb at the recommended levels between 11-12g/dl.

Kidney oxygenation will be evaluated using BOLD-MRI prior to start of therapy, and once again after 24 weeks of treatment with either RD or DA. Primary endpoint is the change in medullary and cortical R2* (inversely proportional to the tissue oxygenation content) after 24 weeks. Secondary endpoints will be albuminuria and urinary levels of ROS (evaluated by electron paramagnetic resonance (EPR) spectroscopy with CPH spin probes).

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes mellitus with anemia caused by DKD, and indication for treatment with erythropoetin/erythropoietin-stimulating drugs.
2. Age 18-75
3. HbA1c >55
4. Diabetes duration 10+ years.
5. Chronic kidney disease (CKD) stage 3-4
6. Symptomatic anemia with Hb <10g/dl
7. Contraception: Female subjects must be postmenopausal, surgically sterile, or if premenopausal (and not surgically sterile), be prepared to use ≥1 effective method of contraception during the study and for 30 days after the last visit. Effective methods of contraception are those listed below:

   1. Double barrier method, i.e. (a) condom (male or female) or (b) diaphragm, with spermicide; or
   2. Intrauterine device; or
   3. Vasectomy (partner); or
   4. Hormonal (e.g., contraceptive pill, patch, intramuscular implant, or injection); or
   5. Abstinence, if in line with the preferred and usual lifestyle of the subject.
8. Signed informed consent.

Exclusion Criteria:

1. Anemia not related to CKD.
2. Dialysis dependent CKD
3. Currently treated for renal anemia using erythropoietin-stimulating drugs
4. Infections during the last 30 days.
5. Severe hypertension (≥180mmHg systolic or >110mmHg diastolic blood pressure)
6. Liver failure (Child-Pugh class B-C)
7. History of epilepsy or seizures
8. Any concomitant disease or condition that may interfere with the possibility for the patient to comply with or complete the study protocol.
9. Ongoing drug or alcohol abuse.
10. Known allergy to RD or DA
11. Malignancy
12. Severe claustrophobia
13. Participation in another ongoing pharmacological study
14. If female: plans to become pregnant, known pregnancy or a positive urine pregnancy test (confirmed by a positive serum pregnancy test), or currently breastfeeding.
15. Unwillingness to participate following oral and written information
16. Other severe acute or chronic medical or psychiatric condition that makes the subject inappropriate for the study, as judged by the investigator.
17. History of thrombosis (DVT, pulmonary embolism)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in kidney oxygenation levels | 24 Weeks
  Kidney oxygenation will be evaluated using BOLD-MRI prior to start of therapy, and once again after 24 weeks of treatment with either RD or DA. Primary endpoint is the change in medullary and cortical R2* (inversely proportional to the tissue oxygenation content) after 24 weeks.

SECONDARY OUTCOMES:
Change in albuminuria | 24 Weeks
  Secondary endpoint will be albuminuria after 24 weeks of either treatment
Change in urinary reactive oxygen species (ROS) | 24 Weeks
  Secondary endpoints will be urinary levels of ROS (evaluated by electron paramagnetic resonance (EPR) spectroscopy with CPH spin probes).

CONTACTS AND LOCATIONS:
Overall Officials: Sergiu Catrina, Ass. Proff., Principal Investigator — Karolinska institute, Centre for diabetes
Locations (1):
- Centre for diabetes, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Catrina SB, Zheng X. Hypoxia and hypoxia-inducible factors in diabetes and its complications. Diabetologia. 2021 Apr;64(4):709-716. doi: 10.1007/s00125-021-05380-z. Epub 2021 Jan 26. PMID 33496820
- [Background] Sebastiani G, Grieco FA, Spagnuolo I, Galleri L, Cataldo D, Dotta F. Increased expression of microRNA miR-326 in type 1 diabetic patients with ongoing islet autoimmunity. Diabetes Metab Res Rev. 2011 Nov;27(8):862-6. doi: 10.1002/dmrr.1262. PMID 22069274
- [Background] Ruiter MS, van Golde JM, Schaper NC, Stehouwer CD, Huijberts MS. Diabetes impairs arteriogenesis in the peripheral circulation: review of molecular mechanisms. Clin Sci (Lond). 2010 Jun 8;119(6):225-38. doi: 10.1042/CS20100082. PMID 20545627
- [Background] Flyvbjerg A. Diabetic angiopathy, the complement system and the tumor necrosis factor superfamily. Nat Rev Endocrinol. 2010 Feb;6(2):94-101. doi: 10.1038/nrendo.2009.266. PMID 20098449
- [Background] Friederich M, Fasching A, Hansell P, Nordquist L, Palm F. Diabetes-induced up-regulation of uncoupling protein-2 results in increased mitochondrial uncoupling in kidney proximal tubular cells. Biochim Biophys Acta. 2008 Jul-Aug;1777(7-8):935-40. doi: 10.1016/j.bbabio.2008.03.030. Epub 2008 Apr 7. PMID 18439413
- [Background] Koyasu S, Kobayashi M, Goto Y, Hiraoka M, Harada H. Regulatory mechanisms of hypoxia-inducible factor 1 activity: Two decades of knowledge. Cancer Sci. 2018 Mar;109(3):560-571. doi: 10.1111/cas.13483. Epub 2018 Jan 27. PMID 29285833
- [Background] Xia X, Lemieux ME, Li W, Carroll JS, Brown M, Liu XS, Kung AL. Integrative analysis of HIF binding and transactivation reveals its role in maintaining histone methylation homeostasis. Proc Natl Acad Sci U S A. 2009 Mar 17;106(11):4260-5. doi: 10.1073/pnas.0810067106. Epub 2009 Mar 2. PMID 19255431
- [Background] Elson DA, Ryan HE, Snow JW, Johnson R, Arbeit JM. Coordinate up-regulation of hypoxia inducible factor (HIF)-1alpha and HIF-1 target genes during multi-stage epidermal carcinogenesis and wound healing. Cancer Res. 2000 Nov 1;60(21):6189-95. PMID 11085544
- [Background] Ceradini DJ, Kulkarni AR, Callaghan MJ, Tepper OM, Bastidas N, Kleinman ME, Capla JM, Galiano RD, Levine JP, Gurtner GC. Progenitor cell trafficking is regulated by hypoxic gradients through HIF-1 induction of SDF-1. Nat Med. 2004 Aug;10(8):858-64. doi: 10.1038/nm1075. Epub 2004 Jul 4. PMID 15235597
- [Background] Catrina SB. Impaired hypoxia-inducible factor (HIF) regulation by hyperglycemia. J Mol Med (Berl). 2014 Oct;92(10):1025-34. doi: 10.1007/s00109-014-1166-x. Epub 2014 Jun 12. PMID 25027070
- [Background] Palm F, Cederberg J, Hansell P, Liss P, Carlsson PO. Reactive oxygen species cause diabetes-induced decrease in renal oxygen tension. Diabetologia. 2003 Aug;46(8):1153-60. doi: 10.1007/s00125-003-1155-z. Epub 2003 Jul 17. PMID 12879251
- [Background] Semenza GL. Pharmacologic Targeting of Hypoxia-Inducible Factors. Annu Rev Pharmacol Toxicol. 2019 Jan 6;59:379-403. doi: 10.1146/annurev-pharmtox-010818-021637. PMID 30625281
- [Background] Pruijm M, Mendichovszky IA, Liss P, Van der Niepen P, Textor SC, Lerman LO, Krediet CTP, Caroli A, Burnier M, Prasad PV. Renal blood oxygenation level-dependent magnetic resonance imaging to measure renal tissue oxygenation: a statement paper and systematic review. Nephrol Dial Transplant. 2018 Sep 1;33(suppl_2):ii22-ii28. doi: 10.1093/ndt/gfy243. PMID 30137579
- See also: Nationella Diabetesregistret 2023 — https://www.ndr.nu/